CLINICAL TRIAL: NCT03183089
Title: A Randomized, Single-Center, Comparative Study of Rohto Dry-Aid® and Systane® Ultra in the Management of Tear Film Stability and Visual Function in Patients With Dry Eye
Brief Title: Comparative Study of Rohto Dry-Aid® and Systane® Ultra in Patients With Dry Eye
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Mentholatum Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-110-0011
Record Dates: First submitted 2017-06-06; First posted 2017-06-09 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Dry Eye Syndromes; Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Experimental)
  Interventions: Drug: Rohto Dry-Aid®
- Active Comparator (Active Comparator)
  Interventions: Drug: Systane® Ultra

INTERVENTIONS:
Drug: Rohto Dry-Aid®
  Arms: Active
Drug: Systane® Ultra
  Arms: Active Comparator

SUMMARY:
The objective of this study is to evaluate the efficacy of Rohto Dry-Aid® in comparison to Systane® Ultra on visual function and tear film stability in patients diagnosed with Dry Eye.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age
* Provide written informed consent
* Have a reported history of dry eye
* Have a history of use of eye drops for dry eye symptoms
* Ocular discomfort
* Conjunctival redness
* Tear film break up time
* Corneal and Conjunctival Staining

Exclusion Criteria:

* Have any clinically significant slit lamp findings at entry visit
* Be diagnosed with an ongoing ocular infection
* Have any planned ocular and/or lid surgeries over the study period
* Have an uncontrolled systemic disease
* Be a woman who is pregnant, nursing or planning a pregnancy
* Be a woman of childbearing potential who is not using an acceptable means of birth control
* Have a known allergy and/or sensitivity to the test article or its components
* Have a condition or be in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-12-03 (Actual); Primary Completion 2016-01-04 (Actual); Study Completion 2016-01-04 (Actual)

PRIMARY OUTCOMES:
Dry Eye Staining | 28 days
  Dry eye syndrome corneal and conjunctival staining assessment
Dry Eye Symptom Questionnaire | 28 days
  Symptom assessment questionnaire
Tear Film Break Up Time | 28 days
  Tear Film Break Up Time after instillation of fluorescein dye
Visual Function Assessment | 28 days
  Reading Test

SECONDARY OUTCOMES:
Drop Comfort Assessment | Day 1
  The comfort of the eye drop will be performed to assess changes from baseline
Visual Acuity | 28 Days
  Visual Acuity will be measured using the EDTRS chart to assess changes from baseline
Slit-Lamp Biomicroscopy | 28 Days
  Slit lamp biomicroscopy exams will be performed to assess any changes from baseline
Adverse Event | 28 Days
  Adverse Event queries

CONTACTS AND LOCATIONS:
Overall Officials: Gail L Torkildsen, M.D., Principal Investigator — Andover Eye Associates
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No